CLINICAL TRIAL: NCT04414748
Title: A Randomized Control Trial to Compare the Euploid Rate of Blastocyst Between the Progestin-primed Ovarian Stimulation Protocol and the GnRH Antagonist Protocol in Patients Undergoing PGT-A
Brief Title: Comparison of the Euploid Rate of Blastocyst Between PPOS and GnRH Antagonist Protocol in Patients Undergoing PGT-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIAI 2020-05
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Preimplantation Genetic Testing; Progestin-primed Ovarian Stimulation; Euploid Rate; GnRH Antagonist
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antagonist group (Active Comparator): Women will receive antagonist (Cetrotide 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.
  Interventions: Drug: GnRH antagonist
- PPOS group (Experimental): Women will receive oral Duphaston 10mg bd from Day 3 till the day of ovulation trigger.
  Interventions: Drug: oral Duphaston

INTERVENTIONS:
Drug: GnRH antagonist — GnRH antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of COH till the day of the ovulation trigger
  Other Names: Cetrorelix
  Arms: Antagonist group
Drug: oral Duphaston — oral Duphaston 10mg bd from Day 3 of COH till the day of ovulation trigger.
  Other Names: Duphaston
  Arms: PPOS group

SUMMARY:
This randomized trial aims to compare the euploid rate of blastocysts between PPOS and GnRH antagonist protocols in patients undergoing PGT-A. Infertile women who have medical indication for PGT-A will be recruited for study after explanation and counseling if they fulfill the inclusion criteria and do not have the exclusion criteria. Eligible women will be randomised into one of the two groups:

Antagonist group: Women will receive antagonist once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.

PPOS group: Women will receive oral Duphaston 10mg bd from Day 3 till the day of ovulation trigger.

The primary outcome is the euploidy rate of blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* Age of women <43 years at the time of ovarian stimulation for IVF
* Antral follicle count (AFC) >=5 on day 2-5 of the period
* PGT-A indicated for advanced maternal age (>=38 years), recurrent miscarriage (>=2 consecutive miscarriage) and repeated implantation failure (>=4 embryos replaced or >=2 blastocysts replaced without success), recurrent foetal aneuploidy

Exclusion Criteria:

* Presence of a functional ovarian cyst with E2>100 pg/mL
* Recipient of oocyte donation
* Presence of hydrosalpinx or endometrial polyp which is not surgically treated

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
euploidy rate | 1 month after oocyte retrieval
  euploidy rate of blastocysts

SECONDARY OUTCOMES:
number of mature oocytes | 1 day after oocyte retrieval
  number of MII oocytes
number and grading of blastocysts | 1 week after oocyte retrieval
  number and grading of blastocysts suitable for biopsy and freezing
positive serum hCG | 2 weeks after FET
  serum β-hCG ≥10 mIU/mL of the first FET
clinical pregnancy | 6 weeks' gestation
  presence of intrauterine gestational sac by trans-vaginal ultrasound at 6 gestational weeks of the first FET
implantation rate | 6 weeks' gestation
  the number of gestational sacs per blastocyst transferred of the first FET
biochemical pregnancy | 6 weeks' gestation
  positive serum hCG not followed by clinical pregnancy of the first FET
ongoing pregnancy | 12 weeks' gestation
  a viable pregnancy beyond 12 weeks' gestation of the first FET
live birth rate | 1 year after FET
  deliveries ≥22 weeks gestation with heartbeat and breath of the first FET
multiple pregnancy | multiple pregnancy beyond gestation 12 weeks
  more than one intrauterine sacs on scanning
ectopic pregnancy | ectopic pregnancy during 12 weeks' gestation
  pregnancy outside the uterine cavity
birthweight of newborns | 1 year after FET
  the birth weight of newborns
serum baseline FSH | day 2-3 of period
  baseline FSH of period day 2-3
progesterone level on the trigger day | 2 days before oocyte retrieval
  progesterone level on the trigger day
estradiol level on the trigger day | 2 days before oocyte retrieval
  estradiol level on the trigger day
miscarriage | 22 weeks of pregnancy
  clinically recognised pregnancy loss before 22 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Study Director — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- Shanghai JiAi Genetics & IVF Institute, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available when beginning 3 months and ending 5 years following article publication.
Access Criteria: To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with. Proposals should be sent to lihe198900@163.com.

REFERENCES:
- [Background] Lee E, Illingworth P, Wilton L, Chambers GM. The clinical effectiveness of preimplantation genetic diagnosis for aneuploidy in all 24 chromosomes (PGD-A): systematic review. Hum Reprod. 2015 Feb;30(2):473-83. doi: 10.1093/humrep/deu303. Epub 2014 Nov 28. PMID 25432917
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Derived] Li H, Yu M, Zhang W, Chen J, Chen H, Lu X, Li L, Ng EHY, Sun X. Comparing blastocyst euploid rates between the progestin-primed and gonadotrophin-releasing hormone antagonist protocols in aneuploidy genetic testing: a randomised trial protocol. BMJ Open. 2024 Mar 23;14(3):e079208. doi: 10.1136/bmjopen-2023-079208. PMID 38521533